CLINICAL TRIAL: NCT04054375
Title: Open Label Safety and Efficacy of Once Weekly Steroid in Patients With LGMD and Becker Muscular Dystrophy
Brief Title: Weekly Steroids in Muscular Dystrophy
Acronym: WSiMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Senda Ajroud-Driss, Associate Professor of Neurology (Neuromuscular Disease), Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00208443
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Limb-girdle Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Steroids, Prednisone
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Duchenne | interventions — Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weekly Steroid (Experimental): Subjects will be asked to take weekly GC oral prednisone dosed based on weight (1mg/kg for patients who weigh less than or equal to 70 kg and 0.75 mg/kg for patients who weigh more than 70 kg). Subjects will also be instructed to take their weekly prednisone on Mondays after their last meal between 7 and 9 PM
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Subjects will be asked to take weekly GC oral prednisone dosed based on weight (1mg/kg for patients who weigh less than or equal to 70 kg and 0.75 mg/kg for patients who weigh more than 70 kg). Subjects will also be instructed to take their weekly prednisone on Mondays after their last meal between 7 and 9 PM
  Other Names: Prednisolone

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of oral weekly glucocorticoid steroids in patients with Becker Muscular Dystrophy (BMD), an inherited disorder in which patients experience weakness of the legs and pelvis, and Limb Girdle Muscular Dystrophy (LGMD), an inherited disorder in which patients experience progressive muscular weakness predominately in their hip and shoulders. The primary objective is safety which we the investigators will measure using laboratory testing and forced vital capacity (FVC), a breathing test that measures the strength of your lungs. The secondary objective is efficacy which will be measured by a change in MRI muscle mass, improved muscle performance, and quality of life.

The investigators hypothesize that patients who receive oral weekly glucocorticoid steroids will have improviements in strength and quality of life compared to their baseline. Furthermore, the investigators anticipate that oral weekly glucocorticoid steroids will not have significant adverse impact on patients.

DETAILED DESCRIPTION:
Glucocorticoid (GC) steroids are a mainstay of therapy for Duchenne Muscular Dystrophy, where they have been shown to prolong ambulation in for DMD in random clinical trials (Gloss et al., 2016). Dosing regimen vary for DMD, but most trials utilized oral daily dosing at 0.75- 1 mg/kg of prednisone or deflazacort (Birnkrant et al., 2018). The age at which to begin oral glucocorticoids and the age at which to cease steroid use are not well established by clinical trial investigation. High dose weekend dosing of oral glucocorticoid steroids has also been suggested to be noninferior to daily dosing when evaluated in a year-long study in DMD, and this approach is preferred in some settings since related to a reduced side effect profile, particularly with respect to behavioral changes which can occur with daily GC steroid dosing in children (Escolar et al., 2011). The use of GC steroids for other forms of muscular dystrophy, including Becker Muscular Dystrophy (BMD) and the Limb Girdle Muscular Dystrophies (LGMDs) is not considered standard of care and has insufficiently been investigated by randomized clinical trials (RCT). An RCT of GC steroids in LGMD 2B (DYSF mutations) was associated with unfavorable outcomes in the steroid treated group (Walter et al., 2013).

Recently, weekly steroid dosing was investigated in preclinical mouse models of muscular dystrophy, including the mdx mouse model of DMD/BMD and two models of LGMD, including LGMD 2B (DYSF) and 2C (SGCG) (Quattrocelli et al., 2017a; Quattrocelli et al., 2017b). All three models showed improved strength and reduced fibrosis with weekly GC steroid dosing. Moreover, in unpublished data, long term studies (24-52 weeks duration) in mice, showed favorable results with improved muscle strength in the mdx and DYSF models.

The investigators propose to carry out an open label safety and efficacy trial of oral weekly GC steroids in patients with BMD and LGMD subtypes. Subjects will be recruited based on age, molecular diagnosis of BMD and LGMD subtypes, and willingness to participate. Both ambulatory and nonambulatory subjects will be included. Subjects will be excluded if they have diabetes mellitus, full time ventilator use, or severely compromised cardiac function, including symptoms referable to heart failure. Subjects must provide consent.

Subjects will be asked to take weekly GC oral prednisone dosed based on weight (1mg/kg for patients who weigh less than or equal to 70 kg and 0.75 mg/kg for patients who weigh more than 70 kg). Subjects will also be instructed to take their weekly prednisone on Mondays after their last meal between 7 and 9 PM. Prior to initiation, subjects will provide a blood sample for baseline screening including serum chemistries, HgbA1-C, creatine kinase, and lipid panel (HDL, LDL, triglycerides, and total cholesterol) and for exploratory biomarkers. Subjects will also provide a urine sample to analyze changes in metabolic biomarkers that are excreted. Subjects will have a physical exam and medical record review. Subjects will have strength testing and complete 10 meter timed run test in addition to a 6 min walk test (if ambulatory). Subjects will be asked to complete quality of life questionnaire. At 6 months, subjects will be evaluated with a physical exam, strength testing, spirometry, 10 meter timed run test and 6 min walk test (if ambulatory), blood draw for serum chemistry, HgbA1-C, creatine kinase, lipid panel and for exploratory biomarkers. Subjects will also provide a urine specimen to be analyzed for any changes in excretion of metabolic markers as an exploratory endpoint. Subjects will be asked to complete a quality of life questionnaire. An MRI/ MRS will be performed before starting GC oral prednisone and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Becker muscular dystrophy or LGMD2A (CAPN3), LGMD 2B (DYSF), LGMD 2C (SGCG), LGMD2E (SGCB), LGMD2F (SGCD), LGMD 2I (FKRP), LGMD (ANO5). Genetic mutation or muscle biopsy staining required to confirm genetic subtype
2. Ages 18-65 years
3. EKG without evidence of prior infarct or atrial fibrillation done within 2 months of study initiation.
4. Echocardiogram with LVEF >25% done within 6 months of study initiation.
5. Stable medications (same medication and dose) for the previous 3 months
6. Stable pulmonary status for the previous 6 months (No change in FVC by more than 20% in the past 6-months)

Exclusion Criteria:

1. Diabetes
2. BMI>35 kg/m2
3. Cardiac transplantation
4. Myocardia Infarct in the past 2-years from screening
5. Any history of tuberculosis
6. Untreated or uncontrolled (medication and/or dose change in previous month from screening) hypertension
7. A diagnosis of congestive heart failure
8. A diagnosis of chronic kidney disease
9. A diagnosis of untreated hypothyroidism
10. The patient is believed to be at high risk of osteoporosis by the primary investigator
11. Inability to provide consent
12. Full time ventilator dependency
13. Heart failure symptoms or LVEF <25%
14. Orthopedic surgery within the prior year or upcoming elective orthopedic surgery within the 6-months from Day 0.
15. Inability to complete MRI (claustrophobia, metal implants)
16. Pregnant women at screening, women seeking to become pregnant, or men seeking to father a child within 6-months from Day 0 should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senda Ajroud-Driss, MD, Principal Investigator — Associate Professor of Neurology (Neuromuscular Disease)
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989
- [Background] Escolar DM, Hache LP, Clemens PR, Cnaan A, McDonald CM, Viswanathan V, Kornberg AJ, Bertorini TE, Nevo Y, Lotze T, Pestronk A, Ryan MM, Monasterio E, Day JW, Zimmerman A, Arrieta A, Henricson E, Mayhew J, Florence J, Hu F, Connolly AM. Randomized, blinded trial of weekend vs daily prednisone in Duchenne muscular dystrophy. Neurology. 2011 Aug 2;77(5):444-52. doi: 10.1212/WNL.0b013e318227b164. Epub 2011 Jul 13. PMID 21753160
- [Background] Gloss D, Moxley RT 3rd, Ashwal S, Oskoui M. Practice guideline update summary: Corticosteroid treatment of Duchenne muscular dystrophy [RETIRED]: Report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2016 Feb 2;86(5):465-72. doi: 10.1212/WNL.0000000000002337. PMID 26833937
- [Background] Quattrocelli M, Barefield DY, Warner JL, Vo AH, Hadhazy M, Earley JU, Demonbreun AR, McNally EM. Intermittent glucocorticoid steroid dosing enhances muscle repair without eliciting muscle atrophy. J Clin Invest. 2017 Jun 1;127(6):2418-2432. doi: 10.1172/JCI91445. Epub 2017 May 8. PMID 28481224
- [Background] Quattrocelli M, Salamone IM, Page PG, Warner JL, Demonbreun AR, McNally EM. Intermittent Glucocorticoid Dosing Improves Muscle Repair and Function in Mice with Limb-Girdle Muscular Dystrophy. Am J Pathol. 2017 Nov;187(11):2520-2535. doi: 10.1016/j.ajpath.2017.07.017. Epub 2017 Aug 18. PMID 28823869
- [Background] Walter MC, Reilich P, Thiele S, Schessl J, Schreiber H, Reiners K, Kress W, Muller-Reible C, Vorgerd M, Urban P, Schrank B, Deschauer M, Schlotter-Weigel B, Kohnen R, Lochmuller H. Treatment of dysferlinopathy with deflazacort: a double-blind, placebo-controlled clinical trial. Orphanet J Rare Dis. 2013 Feb 14;8:26. doi: 10.1186/1750-1172-8-26. PMID 23406536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Diagnosis Subtype:
  19 with Limb-Girdle Muscular Dystrophy
  1 with Becker Muscular Dystrophy
Period: Overall Study
Arm/Group | Weekly Steroid
Started | 20
Completed | 20 (Due to COVID-19, some participants were not able to come to our site to complete all outcome measurements. Our study team worked with individuals to make them feel safe and collect as much data as we possibly could. This is the reason why some outcome metrics have less than 20 data points. All 20 patients completed the study and took the medication for all 24 weeks.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the numbers in the participant flow.
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose
Description: mg/dL, 0-unlimited, higher score indicates worse outcome
Time Frame: Baseline and 6 months (Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 16
mg/dL
  Baseline | 93 (2)
  End | 102 (4)

2. Primary Outcome: HbgA1c
Description: % , 0-100, higher score indicates worse outcome
Time Frame: Baseline and 6 months (Final Visit)
Measure: Mean (Standard Deviation); unit: % A1c
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 17
% A1c
  Baseline | 5.2 (0.08)
  End | 5.3 (0.09)

3. Primary Outcome: Fasting Lipid Profile
Description: cholesterol levels - mg/dL, higher levels indicate worse outcomes
Time Frame: Baseline and 6 months (Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 17
mg/dL
  Baseline | 182 (10)
  End | 185 (9)

4. Primary Outcome: Creatine Kinase
Description: units/L, 0-unlimited, higher scores indicate worse outcome
Time Frame: Baseline and 6 months (Final Visit)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 17
U/L
  Baseline | 1574 (269)
  End | 1047 (171)

5. Primary Outcome: Respiratory Changes
Description: Force Vital Capacity (% of predicted value), decrease in FVC indicates declining respiratory function.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: % Expected
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 11
% Expected
  Baseline | 80 (8)
  End | 79 (8)

6. Secondary Outcome: Functional Assessments - NSAD Change
Description: Northstar Assessment for Dysferlinopathy
  - score out of 58, range from 0 to 58, higher score indicates greater functional ability.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 16
score on a scale
  baseline | 18.4 (17)
  6 months | 18.6 (17)

7. Secondary Outcome: 6 Minute Walk Test
Description: number of meters walked in 6 minute period. Higher values indicate more motor function.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Error); unit: meters
Groups:
- Steroid Group: Participants treated with steroids that were ambulatory.
Arm/Group | Steroid Group
Number analyzed (Participants) | 8
meters
  Baseline | 386 (37)
  6 months | 410 (40)

8. Secondary Outcome: 10 Meter Run Timed
Description: time in seconds to walk/run 10 meters , less time to run indicates greater motor function
Time Frame: Baseline, Month 6
Measure: Mean (Standard Error); unit: seconds
Groups:
- Steroid Treatment: Participants on steroid treatment.
Arm/Group | Steroid Treatment
Number analyzed (Participants) | 9
seconds
  Baseline | 7.32 (0.92)
  6 months | 6.67 (0.77)

9. Secondary Outcome: Brooke Scale Score
Description: upper extremity assessment, scoring between 1- 6, lower score indicates more upper extremity function
Time Frame: Baseline, Month 6
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 18
scores on a scale
  baseline | 3 (1)
  6 months | 3 (1)

10. Secondary Outcome: Vignos Scale Score
Description: Lower extremity assessment, score from 1-10, lower score indicates more function.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Steroid Treatment Group: Participants treated with steroids
Arm/Group | Steroid Treatment Group
Number analyzed (Participants) | 20
scores on a scale
  baseline | 5 (1)
  6 months | 5 (1)

11. Secondary Outcome: Muscle Imaging
Description: MRI of leg muscles to measure changes in muscle fat percentage. The data point was collected by taking fat percentage at 6 months minus fat percentage at baseline with the following equation: (([final fat percentage - initial fat percentage]/initial fat percentage) * 100%)). All participants were included, both ambulatory and nonambulatory, with all genetic subtypes included. Five participants didn't have an MRI scan at 6 months and therefore were not included. Muscles imaged were analyzed for muscle fat changes from baseline to 6 months. Data is limited in interpretation due to various muscle groups in both ambulatory and non-ambulatory patients.
Time Frame: Baseline, 6 months
Population: MRI of the muscles was collected on all baseline patients (20 participants). Due to clinical heterogeneity, different muscles had to be imaged for each patient. Five participants didn't get follow-up MRI scans due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: percent of change from baseline
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 15
percent of change from baseline | -14 (13)

12. Secondary Outcome: Bone Density
Description: whole dexa body scan to assess bone density with Z scores (more negative z score indicates increased risk for fractures).
  Z-score of 0 represents the population mean, and is the average bone density. Positive scores indicate greater bone density and negative scores indicate decreased bone density, which could be clinically correlated with osteoporosis.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 15
z-score
  baseline | -1.64 (0.33)
  6 months | -1.65 (0.34)

13. Secondary Outcome: Lean Mass %
Description: whole body dexa scans to assess lean mass % (0- 100 %). Increase lean mass % is the desired outcome.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 15
percentage
  baseline | 37.5 (2.5)
  6 months | 38.1 (2.6)

14. Secondary Outcome: Functional Assessments - Upper Limb Strength
Description: Grip strength of the total force (Newtons) in both hands.
  Participants attempted 3 trials in the right hand that was then averaged to create a right-hand average force score.
  Then, the participants attempted 3 trials in the left hand that was then averaged to create a left-hand average force score.
  The right-hand average force score was added to the left-hand average force score to create a total grip strength score.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Force (Newtons)
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 17
Force (Newtons)
  Baseline | 39 (25)
  6 months | 41 (27)

15. Secondary Outcome: Muscle Strength Test
Description: Manual motor testing of the right knee flexion muscle group.
Time Frame: baseline, 6 months
Population: Manual muscle testing scores are from 0 to 5, with 5 being the strongest and 0 no muscle movement at all.
Measure: Mean (Full Range); unit: Units on scale
Arm/Group | Weekly Steroid
Number analyzed (Participants) | 16
Units on scale
  Baseline | 3 [1 to 5]
  6 months | 3 [1 to 5]

ADVERSE EVENTS:
Time Frame: Participants were monitored for 24 weeks or 6 months while taking study drug.
Arm/Group | Weekly Steroid
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Some patients were not able to complete the study visits at end of the study due to COVID-19 and fearing safely coming to our site for visits. This is why many metrics do not have 20 data points. All patients completed the 24 weeks of steroid dosing and adverse event check-in. No participants left the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04054375/Prot_001.pdf